CLINICAL TRIAL: NCT05543057
Title: Real-world Study on Comprehensive Treatment of Esophageal Cancer Based on Precision Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zefen Xiao (Unknown)
Responsible Party: Sponsor-Investigator, Zefen Xiao, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: 22/036-3237
Record Dates: First submitted 2022-09-08; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Esophageal Cancer
Keywords: Real-world study; Individualized regimen; Liquid biopsy; Prediction models
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — The blood and saliva samples before, during and after radiotherapy; the remaining diagnostic biopsy tissue samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: 3DCRT — Three-dimensional conformal radiotherapy (3DCRT)

SUMMARY:
Radiotherapy is one of the main treatments for locally advanced esophageal carcinoma (EC). The accuracy of the existing imaging methods in diagnosing and predicting therapeutic efficacy is disappointing, which increases the difficulty in clinical decision-making. In this study, based on a continuous cohort of EC treated with radiotherapy, the clinical and pathological factors of the patients are used to classify them into the appropriate therapeutic group. By multiple liquid biopsy technologies, combining with radiomics, we intend to construct prediction models of prognosis, therapeutic effect and toxicity. The aim of this RWS is to provide appropriate individualized regimen, further optimize the treatment mode based on precision radiotherapy and improve the outcome and quality of life of EC patients.

DETAILED DESCRIPTION:
Radiotherapy is one of the main treatments for locally advanced esophageal squamous cell carcinoma (ESCC). The guidelines recommend neoadjuvant concurrent chemoradiotherapy plus surgery for resectable or potentially resectable patients; for unresectable patients, definitive chemoradiotherapy is the standard treatment. However, due to the complexity of the biological behavior of esophageal cancer (EC) and individual differences, fully complying with guideline recommendations in clinical practice is difficult and idealized. The results of prospective clinical trials are difficult to meet the demand of clinical diagnosis and treatment, thus, carrying out high-quality real-world study (RWS) is necessary.

Three-dimensional conformal radiotherapy (3DCRT) for unresectable EC yields 5-year OS rates of 34%-45.6%, which is an improvement over the rates reported in the RTOG 85-01 and 94-05 studies. Even so, there is still room for improvement of local control rate and overall survival. The accuracy of the existing imaging methods [computed tomography (CT), magnetic resonance imaging (MRI), endoscopic ultrasonography (EUS), endoscopic ultrasonography (EUS), as well as positron-emission tomography (PET)-CT, etc.] in diagnosing and predicting therapeutic efficacy is disappointing, which increases the difficulty in clinical decision-making. It is worthy to investigate an appropriate individualized radiation regimen based on different treatment sensitivity.

In this study, based on a continuous cohort of EC treated with radiotherapy, the clinical and pathological factors of the patients are used to classify them into the appropriate therapeutic group. Collect the blood and saliva samples before, during and after radiotherapy; the remaining diagnostic biopsy tissue samples. By using multiple liquid biopsy technologies [microbial flora, circulating tumor DNA (ctDNA), genome, RNA, and immunophenotype, ect.], combining with radiomics, construct prediction models of prognosis, therapeutic effect and toxicity. The aim of this RWS is to provide appropriate individualized regimen, further optimize the treatment mode based on precision radiotherapy and improve the outcome and quality of life of EC patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathology proved esophageal cancer
* ECOG PS ≤3
* Signed Informed consent

Exclusion Criteria:

* Pregnant and lactating women
* Others that researchers consider inappropriate

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer who are acceptable and tolerable to radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
1-, 2-, 3-year overall survival | From treatment initiation to death from any cause or censor, assessed up to 36 months
  Overall survival

SECONDARY OUTCOMES:
1-, 2-, 3-year progression-free survival | From treatment initiation to first documented progression or death or censor, assessed up to 36 months
  Progression-free survival
Rate of acute toxicity (any and above grade 3) | From enrollment to 3 months after treatment
  Toxicities according to CTCAE criteria
Rate of acute/late toxicity (any and above grade 3) | After 3 months of enrollment
  Toxicities of chemoradiation therapy
1-month short-term efficacy | Assessed 1-month after radiotherapy (short-term) according to RECIST 1.1
  Short-term efficacy
Quality of Life change, QoL | 1/3/6/12/24 months after radiotherapy
  measurement basing on EORTC (Quality of life of patients with oesophageal cancer) QLQ-C30 tables
Quality of life of patients with oesophageal cancer | 1/3/6/12/24 months after radiotherapy
  measurement basing on EORTC (Quality of life of patients with oesophageal cancer) QLQ-OES18 tables

OTHER OUTCOMES:
Biomarkers to predict radiotherapy efficacy | baseline/through study completion, an average of 2 year
  potential biomarkers in tumor samples and blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, Beijing Municipality, China